CLINICAL TRIAL: NCT05633810
Title: COLchicine and Non-enteric Coated Aspirin in the Cardiovascular Outcomes Trial of Patients With Type 2 Diabetes (COLCOT-T2D)
Brief Title: COLchicine and Non-enteric Coated Aspirin in the Cardiovascular Outcomes Trial of Patients With Type 2 Diabetes
Acronym: COLCOT-T2D
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MHICC-2021-001
Record Dates: First submitted 2022-11-11; First posted 2022-12-01 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Diabete Type 2; Cardiovascular Diseases
Keywords: Diabetes (Type 2); Heart Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Heart Diseases | interventions — Aspirin; Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Anti-thrombotic arm (Active Comparator): For patients eligible for aspirin therapy arm.
  Interventions: Drug: Aspirin; Drug: Aspirin Placebo; Drug: Colchicine; Drug: Colchicine Placebo
- Anti-thrombotic arm (Placebo) (Placebo Comparator): For patients eligible for aspirin therapy arm.
  Interventions: Drug: Aspirin; Drug: Aspirin Placebo; Drug: Colchicine; Drug: Colchicine Placebo
- Anti-inflammatory arm (Active Comparator): For patients ineligible for aspirin therapy arm.
  Interventions: Drug: Colchicine; Drug: Colchicine Placebo
- Anti-inflammatory arm (Placebo) (Placebo Comparator): For patients ineligible for aspirin therapy arm.
  Interventions: Drug: Colchicine; Drug: Colchicine Placebo

INTERVENTIONS:
Drug: Aspirin — 40 mg non-enteric-coated tablet taken twice daily.
  Arms: Anti-thrombotic arm; Anti-thrombotic arm (Placebo)
Drug: Aspirin Placebo — non-enteric-coated tablet taken twice daily.
  Arms: Anti-thrombotic arm; Anti-thrombotic arm (Placebo)
Drug: Colchicine — 0.5 mg tablet taken once daily
Drug: Colchicine Placebo — tablet taken once daily.

SUMMARY:
To evaluate the efficacy and safety of colchicine and non-enteric coated aspirin, combined or alone, to improve cardiovascular outcomes in high-risk patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 55 to 80 years
2. Type 2 diabetes treated as per national guidelines
3. No previous history of coronary artery disease-related clinical event
4. And at least one of the following:

   1. Duration of diabetes of 5 years or more,
   2. HbA1c ≥ 8.0% or more in the last 2 years
   3. Active cigarette smoking,
   4. High hs-CRP (> 2.0 mg/L),
   5. High coronary calcium score (Agatston score >100),
   6. High TG-levels (≥1.7 mmol/L) despite lipid lowering therapy administered as per guidelines,
   7. High LDL-C levels (≥3.5 mmol/L) or high non-HDL-C levels (≥4.2 mmol/L) despite lipid lowering therapy administered as per guidelines
   8. High Apo-B (≥1.05 g/L)
   9. Reduced HDL-C (<1.05 mmol/L in men, <1.3 mmol/L in women),
   10. Lp(a) >50 mg/dL,
   11. Peripheral artery disease with stenosis ≥50% or prior revascularization,
   12. Cerebrovascular disease with stenosis ≥50% or prior revascularization,
   13. Diabetic retinopathy or diabetic neuropathy,
   14. Mild or moderate proteinuria (dipstick analysis) or micro-albuminuria
5. Women of childbearing potential must have a negative urine pregnancy test at screening/randomization visit 1 and must agree to use an effective method of birth control throughout the study. Acceptable means of birth control include: oral contraceptives, implantable contraceptives, injectable contraceptives, transdermal contraceptives, intrauterine devices, male or female condoms with spermicide, abstinence, or a sterile sexual partner.

   Women are considered not of childbearing potential if they either:
   1. Have had a hysterectomy or tubal ligation prior to baseline visit or
   2. Are postmenopausal defined as no menses for 12 months or a FSH level (if available) in the menopausal range.
6. Patients with the capacity to provide informed consent.

Exclusion Criteria:

1. Any prior history of myocardial infarction, angina, coronary revascularization, coronary stenosis >30%, stroke, transient ischemic attack, or known heart failure
2. Known chronic renal insufficiency defined as an estimated glomerular filtration rate (eGFR), using the MDRD equation, of < 35 mL/min/1.73m2
3. History of cancer or lymphoproliferative disease within the last 3 years other than a successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix and/or low-grade prostate cancer
4. Inflammatory bowel disease (Crohn's disease or ulcerative colitis) or chronic diarrhea
5. Peptic ulcer diagnosed within the last 24 months or previous gastro-intestinal bleeding, except for mild hemorrhoidal bleeding more than 5 years ago which is permitted (patients meeting this exclusion criterion will not be randomized to receive aspirin or placebo but can be randomized to receive colchicine or placebo)
6. Pre-existent progressive neuromuscular disease or known CPK level > 3 times the upper limit of normal as measured within the past 30 days and determined to be non-transient through repeat testing
7. Any of the following known parameters as measured within the past 90 days, and determined to be non-transient through repeat testing:

   1. hemoglobin < 100 g/L
   2. 2. white blood cell count < 3.0 X 10⁹/L
   3. platelet count <110 X 10⁹/L
   4. ALT > 3 times the upper limit of normal (ULN)
   5. total bilirubin > 2 times ULN (unless due to Gilbert syndrome, which is allowed)
8. History of cirrhosis, chronic active hepatitis or severe hepatic disease
9. Female patient who is pregnant, or breast-feeding or is considering becoming pregnant during the study or for 6 months after the last dose of study medication
10. History of clinically significant drug or alcohol abuse in the last year
11. Patient is currently using or plans to begin chronic systemic steroid therapy (oral or intravenous) during the study (topical or inhaled steroids are allowed, as well as replacement corticosteroids for adrenal insufficiency)
12. Current chronic treatment with aspirin or another antiplatelet agent (patients meeting this exclusion criterion will not be randomized to receive aspirin or placebo but can be randomized to receive colchicine or placebo)
13. Chronic treatment with an anticoagulant agent (patients meeting this exclusion criterion will not be randomized to receive aspirin or placebo but can be randomized to receive colchicine or placebo)
14. Current use of colchicine for other indications (mainly chronic indications consisting of Familial Mediterranean Fever or gout); there is no wash-out period required for patients who have been treated with colchicine and stopped treatment prior to enrolment
15. History of an allergic reaction or significant sensitivity to colchicine
16. History of an allergic reaction or significant sensitivity to aspirin (patients meeting this exclusion criterion will not be randomized to receive aspirin or placebo but can be randomized to receive colchicine or placebo)
17. Chronic treatment with an anti-inflammatory agent (for example, anti-TNF-alpha or nonsteroidal anti-inflammatory drug (NSAID))
18. Use of an investigational chemical agent less than 30 days or 5 half-lives prior to the screening visit (whichever is longer)
19. Patient is considered by the investigator, for any reason, to be an unsuitable candidate for the study.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2022-12-21 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
First event of the composite of cardiovascular death, resuscitated cardiac arrest, non-fatal myocardial infarction, non-fatal stroke, or urgent hospitalization for angina requiring coronary revascularization. | From randomization to occurrence of first event, assessed up to 60 months.
  The number of participants having at least one of the composite of the primary endpoint.

SECONDARY OUTCOMES:
Cardiovascular Death | From randomization to cardiovascular death, assessed up to 60 months.
  The number of participants having a cardiovascular death.
First Event of Resuscitated Cardiac Arrest | From randomization to event, assessed up to 60 months.
  The number of participants having at least 1 resuscitated cardiac arrest.
First Event of Non-fatal Myocardial Infarction | From randomization to event, assessed up to 60 months.
  The number of participants having at least 1 myocardial infarction.
First Event of Non-fatal Stroke | From randomization to event, assessed up to 60 months
  The number of participants having at least 1 stroke.
First Occurrence of Urgent Hospitalization for Angina Requiring Coronary Revascularization | From randomization to occurrence, assessed up to 60 months.
  The number of participants having at least 1 urgent hospitalization for angina requiring coronary revascularization.
First Event of Atrial Fibrillation | From randomization to event, assessed up to 60 months.
  The number of participants having at least 1 atrial fibrillation.
First Occurrence of Heart Failure Hospitalization | From randomization to occurrence, assessed up to 60 months.
  The number of participants having at least 1 heart failure hospitalization.
First Occurrence of Coronary Revascularization | From randomization to occurrence, assessed up to 60 months.
  The number of participants having at least 1 coronary revascularization.
MoCA Scores Assessed Over Time | From randomization to yearly follow-ups until the end-of-study visit, assessed up to 60 months.
  Change from randomization in MoCA score at yearly follow-ups (excluding the first-year visit) until the end-of-study visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No